CLINICAL TRIAL: NCT00229684
Title: A 24-week, Randomised, Parallel-Group, Multi-Centre, Open-Label Study of the Renal Effects of Tesaglitazar in Patients With Type 2 Diabetes Mellitus
Brief Title: ARMOR (Analyzing Renal Mechanisms of Creatinine Excretion in Patients On tesaglitazaR)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The development program has been terminated
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: D6160C00040
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — tesaglitazar; Pioglitazone

INTERVENTIONS:
Drug: Tesaglitazar — 2 mg once daily in oral form
  Other Names: Galida
Drug: pioglitazone — 45 mg once daily in oral form
  Other Names: Actos

SUMMARY:
This is a prospective 24-week, randomized, parallel-group, multi-center, active-controlled (pioglitazone 45 mg) open-label study designed to assess the effects of tesaglitazar 2 mg per day on components of renal excretion of creatinine in type 2 diabetics. The study comprises a 2-week enrollment period, followed by a 24-week double blind treatment period and an 8-week follow-up period

ELIGIBILITY:
Inclusion Criteria:

* Provision of a written informed consent
* Men or women who are >=45 years of age
* Female patients: postmenopausal, hysterectomized, or if of childbearing potential, using a reliable method of birth control
* Diagnosed with type 2 diabetes
* Treated with diet alone or treatment with a single oral antidiabetic agent or low doses of two oral antidiabetic agents

Exclusion Criteria:

* Type 1 diabetes
* New York Heart Association heart failure Class III or IV
* Treatment with chronic insulin
* History of hypersensitivity or intolerance to any peroxisome proliferator-activated receptor agonist (like Actos or Avandia), fenofibrate, metformin or 3-hydroxy-3-methylglutaryl coenzyme A reductase inhibitor (statin)
* History of drug-induced myopathy or drug-induced creatine kinase elevation, liver enzyme elevations, neutropenia (low white blood cells)
* Creatinine levels above twice the normal range
* Creatine kinase above 3 times the upper limit of normal
* Received any investigational product in other clinical studies within 12 weeks
* Any clinically significant abnormality identified on physical examination, laboratory tests or electrocardiogram, which in the judgment of the investigator would compromise the patient's safety or successful participation in the clinical study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-09; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Effects of on tubular secretion of creatinine in type 2 diabetics after 12 weeks of treatment as assessed through determinations of:
Glomerular filtration rate (GFR) by iothalamate clearance
Endogenous creatinine clearance

SECONDARY OUTCOMES:
Effects of on tubular secretion of creatinine in type 2 diabetics after 24 weeks of treatment as assessed through determinations of:
GFR by iothalamate clearance
Endogenous creatinine clearance
The time course of change in serum creatinine concentration and GFR during a 24-week period of tesaglitazar treatment in type 2 diabetics
The effects of tesaglitazar on urinary protein excretion in type 2 diabetics by comparisons of urinary total protein and albumin excretion rates
The effects of tesaglitazar on urinary creatinine excretion in type 2 diabetics by comparisons of urinary total creatinine excretion rates
The pharmacokinetics of tesaglitazar during 24 weeks of therapy in type 2 diabetics.
The safety and tolerability of tesaglitazar in type 2 diabetics by assessments of adverse events, laboratory values, electrocardiogram, pulse, blood pressure, body weight, and physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Galida Medical Science Director, MD, Study Director — AstraZeneca
Locations (21):
- United States (21):
  - Research Site, Pasadena, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Gainesville, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site, New Orleans, Louisiana
  - Research Site, Reno, Nevada
  - Research Site, Flushing, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Tulsa, Oklahoma
  - Research Site, Cheswick, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Midland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Gig Harbor, Washington
  - Research Site, Seattle, Washington